CLINICAL TRIAL: NCT07388784
Title: Exploration of the Functional Effect of Modified Gain Precalculation on Soft Speech Intelligibility
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sebastian Griepentrog (Industry)
Responsible Party: Sponsor-Investigator, Sebastian Griepentrog, Clinical studies manager, Sonova AG
Organization: Sonova AG (Industry)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: SRF-35145
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Hearing Loss
MeSH Terms: conditions — Hearing Loss | interventions — Hearing Aids

STUDY DESIGN:
Intervention Model Description: Each participant will be treated with each gain precalculation principle in a randomized order
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Competitor device, hearing aid with standard gain precalculation principle (Active Comparator): Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The active comparator condition is the state of the art hearing aid gain precalculation from a competitor device.
  Interventions: Device: Hearing aid with gain precalculation principle 1; Device: Hearing aid with gain precalculation principle 2
- Hearing aid with gain precalculation principle 1 (Experimental): Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The experimental conditions vary in their parametrization to result in different degrees of added amplification.
  Interventions: Device: Competitor device, hearing aid with standard gain precalculation principle
- Hearing aid with gain precalculation principle 2 (Experimental): Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The experimental conditions vary in their parametrization to result in different degrees of added amplification.
  Interventions: Device: Competitor device, hearing aid with standard gain precalculation principle

INTERVENTIONS:
Device: Competitor device, hearing aid with standard gain precalculation principle — Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The active comparator condition is the state of the art hearing aid gain precalculation from a competitor device.
  Arms: Hearing aid with gain precalculation principle 1; Hearing aid with gain precalculation principle 2
Device: Hearing aid with gain precalculation principle 1 — Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The experimental conditions vary in their parametrization to result in different degrees of added amplification.
  Arms: Competitor device, hearing aid with standard gain precalculation principle
Device: Hearing aid with gain precalculation principle 2 — Each participant will be fitted with two different pairs of hearing aids with different gain precalculation principles. Gain precalculation applies the amplification of sound signals in the hearing aid. The experimental conditions vary in their parametrization to result in different degrees of added amplification.
  Arms: Competitor device, hearing aid with standard gain precalculation principle

SUMMARY:
An exploratory investigation of gain precalculation principles in CE-labelled Sonova brand hearing instruments (e.g. Phonak hearing instruments) is intended to be conducted on hearing impaired participants. These gain precalculation principles are enabled by respective hearing instrument technologies and hearing instrument algorithms. The aim of the study is to investigate and assess strength and weaknesses of these gain precalculation principles in terms of speech intelligibility to determine their application in hearing instruments (Phase of development). Objective laboratory measurements as well as subjective ratings will be carried out. This will be a controlled, single blinded and randomized active comparator clinical evaluation which will be conducted mono centric at Sonova AG Headquarter based in Stäfa.

ELIGIBILITY:
Inclusion Criteria:

* Hearing impaired adult at a minimum age of 18 years
* Good written and spoken german skills
* Ability to fill in a questionnaire concientiously
* Ability to produce a reliable hearing test result
* Ability to describe listening impressions / experiences
* Audiogram is in the fitting range of the hearing aids

Exclusion Criteria:

* Unaidable hearing loss in one or both ears
* Auricle deformities that prevent secure placement of the investigational device
* Acute tinnitus in one or both ears
* Unwillingness to test the investigational device
* Asymmetrical hearing loss
* Hypersensitivity or allergy against synthetic materials
* Symptoms of vertigo or dizziness
* Suffering from any otologic disease

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Estimated)
Dates: Start 2026-03-20 (Estimated); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Speech intelligibility | From enrollment to the end of treatment at 3 weeks
  Speech intelligibility in % will be assessed with a monosyllabic word recognition test for each of the interventional conditions

SECONDARY OUTCOMES:
Qualitative ratings on naturalness | From enrollment to the end of treatment at 3 weeks
  Sound Signals will be rated in terms of naturalness on a scale from 0 - 100 in increments of 1 for each interventional condition
Qualitative ratings on loudness | From enrollment to the end of treatment at 3 weeks
  Sound Signals will be rated in terms of perceived loudness on a scale from 1 - 5 in increments of 1 for each interventional condition
Qualitative ratings on own voice quality | From enrollment to the end of treatment at 3 weeks
  Own voice will be rated in terms of perceived bothersomeness on a scale from 1 - 5 in increments of 1 for each interventional condition

CONTACTS AND LOCATIONS:
Overall Officials: Josephine Hollenbach, Principal Investigator — Sonova AG
Locations (1):
- Sonova AG, Stäfa, Switzerland

IPD SHARING:
Plan to Share IPD: No